CLINICAL TRIAL: NCT04647851
Title: Effects of a Remote Exercise Intervention on Aerobic Endurance, Strength, Gait and Balance in Individuals With Down Syndrome - Pilot Study
Brief Title: Remote Exercise Study for Individuals With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Thessa Hilgenkamp, Assistant Professor, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1442844Pilot
Record Dates: First submitted 2020-11-24; First posted 2020-12-01 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Pre- and post test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote exercise intervention Down syndrome (Experimental): Intervention: The program we will be using is specifically developed for individuals with Down syndrome based on the Mann Method PT Principles. The MMPT Principles TM focus on a progressive program of therapeutic activity (cardiovascular activity), therapeutic exercise (foundational strengthening and hip strengthening activities), and neuromuscular rehabilitation (visual/vestibular and balance activities) to address the unique needs of individuals with Down syndrome. This program has been developed and successfully implemented in Down syndrome activity centers across the country. This program will be offered through Zoom. Intensity will be submaximal for both data collection and during the exercise sessions, and recorded with Polar heart rate monitors.
  Interventions: Other: Remote exercise intervention Down syndrome

INTERVENTIONS:
Other: Remote exercise intervention Down syndrome — See arm description

SUMMARY:
This pilot study aims to test whether remote delivery of the exercise intervention provides a sufficient training stimulus. This pilot study will be remote and online-only, and will have no in-person interaction, data collection or intervention. 20 Participants will participate in a 12-wk, 3hrs/wk remote exercise intervention and in a pre- and a posttest remote testing session. We will use Zoom for all testing and exercise sessions.

DETAILED DESCRIPTION:
Design: Repeated measures design: 20 participants will participate in the remote exercise intervention study with a pre-test and a post-test to investigate training effects on aerobic endurance, strength, balance and gait.

Intervention: The program we will be using is specifically developed for individuals with Down syndrome based on the Mann Method PT Principles. The MMPT Principles TM focus on a progressive program of therapeutic activity (cardiovascular activity), therapeutic exercise (foundational strengthening and hip strengthening activities), and neuromuscular rehabilitation (visual/vestibular and balance activities) to address the unique needs of individuals with Down syndrome. This program has been developed and successfully implemented in Down syndrome activity centers across the country. This program will be offered through Zoom. Intensity will be submaximal for both data collection and during the exercise sessions, and recorded with Polar heart rate monitors.

Measurements: We will use only field tests instead of the original lab-based testing for aerobic endurance, strength, balance and gait, and all tests will be conducted remotely.

Baseline measurements: height, weight, circumferences Aerobic endurance: 2 Minute Step Test: participant marches in place as fast as possible with a set height for how high to lift the knees, for two minutes. Outcome is heart rate and number of steps in two minutes.

Strength: 30 Second Chair Stand and 5 Times Chair Stand: participants starts seated, then stands up and sits down as fast as possible, first counting the number of times within 30 seconds, then timing the number of seconds for 5 times.

Balance: Timed Up and Go: This is a timed test where the participant stands up from a chair, walk 10ft, turn around, walk back and sit down again, as fast as possible. Modified CTSIB (Clinical Test on Sensory Information on Balance) and FICSIT-4 (Frailty and Injuries: Cooperative Studies of Intervention Techniques): Standing balance in different conditions and positions. Functional Reach Test: Reaching from a standing position as far as possible.

Gait: Comfortable and Fast Walking Speed, Observational Gait Analysis based on anterior, posterior and lateral video recordings of the participant's walking.

Additionally, participants (and/or parents/caregivers for the group with Down syndrome) will complete a health history questionnaire and physical activity questionnaire, a questionnaire about risk of falling (Short Falls Efficacy Scale-1) and about attitudes towards exercise (Health Matters Evaluation Toolkit).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years old
* generally healthy
* sedentary (defined as being involved in less than 30 minutes of moderately-intense physical activity per day)
* additionally for the participants with Down syndrome:

  * diagnosis of Down syndrome trisomy 21 and
  * normal thyroid function or stable thyroid function (and medications) for at least 6 mo.

Exclusion Criteria:

* congenital heart disease;
* atherosclerotic or other vascular disease;
* asthma or other pulmonary disease;
* hypertension (defined BP >140/90 mmHg);
* blood pressure below 90/60 mmHg;
* history of pre-syncope or syncope;
* diabetes (defined as Hba1c of >7.5% or use of glucose lowering medication);
* severe obesity (defined as BMI >40);
* medications affecting heart rate, blood pressure or arterial function;
* anti-inflammatory medication including NSAIDS;
* current smoking and
* pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Aerobic endurance | 13 weeks
  We measure aerobic endurance with the 2-min Step Test, outcome measure is number of times the right leg is lifted.

SECONDARY OUTCOMES:
Leg strength | 13 weeks
  30 Second Chair Stand, measured in number of times to stand up.
Leg strength | 13 weeks
  5 times Chair Stand, measured in number of seconds it takes to stand up and sit down 5 times.
Balance | 13 weeks
  Timed Up and Go, measured in seconds to complete task.
Balance | 13 weeks
  Modified CTSIB (Clinical Test on Sensory Information on Balance), measured in seconds
Balance | 13 weeks
  FICSIT-4 (Frailty and Injuries: Cooperative Studies of Intervention Techniques, measured in seconds
Balance | 13 weeks
  Functional reach, measured in centimeter
Gait | 13 weeks
  Walking speed, measured in meter/second
Gait | 13 weeks
  Observational Gait Analysis, measured in total score for deviations

CONTACTS AND LOCATIONS:
Overall Officials: Thessa Hilgenkamp, Ph.D, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual patient data will be made available to other researchers upon request.

REFERENCES:
- [Derived] Hilgenkamp T, Lum R, Roys C, Souza T, Stopka D, Mann S, Ho KY. Effects of a 12-week telehealth exercise intervention on gait speed and gait deviations in adults with Down syndrome. J Intellect Disabil Res. 2024 Jun;68(6):598-609. doi: 10.1111/jir.13132. Epub 2024 Mar 13. PMID 38481070
- [Derived] Guerrero K, Umagat A, Barton M, Martinez A, Ho KY, Mann S, Hilgenkamp T. The effect of a telehealth exercise intervention on balance in adults with Down syndrome. J Appl Res Intellect Disabil. 2023 Mar;36(2):385-393. doi: 10.1111/jar.13068. Epub 2022 Dec 30. PMID 36585748